CLINICAL TRIAL: NCT05185596
Title: Feasibility of Prehospital Trans Esophageal Echocardiography in Cardiac Arrest
Brief Title: Prehospital TEE in Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Berufsrettung Wien (Unknown)
Responsible Party: Principal Investigator, Thomas Hamp, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17182019
Record Dates: First submitted 2021-12-08; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Echocardiography, Transesophageal; Out-of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trans-esophageal echocardiography (Experimental): Transesophageal Echocardiography during advanced life support for out of hospital cardiac arrest will be performed.
  Interventions: Device: Transesophageal Echocardiography

INTERVENTIONS:
Device: Transesophageal Echocardiography — transesophageal Echocardiography during advanced life support

SUMMARY:
This study shall investigate the feasibility of prehospital performed trans-esophageal echocardiography in out of hospital cardiac arrest.

The investigators will include ten patients undergoing advanced life support in this study and determine if it is possible to acquire adequate trans-esophageal images within 10 minutes after arrival of the study team on scene.

DETAILED DESCRIPTION:
Out of hospital cardiac arrest (OOHCA) remains a leading cause of death in Austria.

Current guidelines recommend to address potentially reversible causes for OOHCA early to improve survival and some of these causes can be recognized using echocardiography. The usefulness of trans-thoracic echocardiography during OOHCA seems to be limited as image acquisition may prolong now flow time and image quality is variable. These limitations might be overcome with trans-esophageal echocardiography.

The investigators will investigate the feasibility of prehospital performed trans-esophageal echocardiography in ten OOHCA patients undergoing advanced life support.

In addition to routine care by paramedics and emergency physicians, a dedicated expert in emergency ultrasound will perform trans-esophageal echocardiography in these patients.

Primary outcome parameter: Is it possible to obtain trans-esophageal images of the heart within 10 minutes after arrival of the study team?

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing advanced life support for out of hospital cardiac arrest

Exclusion Criteria:

* patients who should undergo rapid transport to the hospital with ongoing CPR (ECMO candidates, pregnant, trauma, obvious reversible which can be treated in hospital only)
* known esophageal pathology contraindicating TEE
* no definite secure airway present (endotracheal intubation, tracheostomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-11 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to obtain images of the heart | 10 minutes
  Time from arrival of the study team on scene, until the following questions are answered by trans esophageal echocardiography: "is spontaneous cardiac movement present", "how ist LV function", "how is RV function", "is a pericardial effusion or tamponade present". The time will be measured in seconds and a maximum of 600 seconds is allowed. If answering the questions within 600 seconds is possible, the case will be counted as "feasible" and the duration of the time measured will be recorded. If answering the questions takes longer than 10 minutes, the case will be counted as "not feasible"

SECONDARY OUTCOMES:
Hands off times | 10 minutes
  what are the "hands off times" (defined as time during which no chest compressions are performed during the resuscitation) during ALS with or without TEE.
Hindering of advanced life support measures | 10 minutes
  The number of events that hinder the established advanced life support measures will be counted graded by severity (minimal, minor, major)
Trans esophageal echocardiography related complications | 10 minutes
  What complications are caused by trans esophageal echocardiography occur during ALS: displacement of the endotracheal tube, dental injury, pharyngeal injury
Image quality | 10 minutes
  How is image quality of trans esophageal echocardiography during advanced life support measures? This will be determined by the investigator performing the trans esophageal echocardiography and also by a blinded specialist afterwards. The rating will be "excellent", "good", "moderate", "poor", "extremely poor"

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hamp, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No